CLINICAL TRIAL: NCT02063932
Title: Association Between Confocal Laser Endomicroscopic (CLE) Features and Gastric Mucosal Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2014SDU-QILU-G02
Record Dates: First submitted 2014-01-29; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Mucosal Microbiome; H.Pylori; Intestinal Metaplasia; Gastric Neoplasia
Keywords: mucosal microbiome; H.pylori; intestinal metaplasia; gastric neoplasia; endomicroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The metagenome was obtained from biopsy specimen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- endomicroscopy
  Interventions: Other: endomicroscopy, targeted biopsy and 16s rRNA gene sequencing

INTERVENTIONS:
Other: endomicroscopy, targeted biopsy and 16s rRNA gene sequencing

SUMMARY:
There might be a correlation between gastric mucosal microbiome and mucosal pattern visualized by confocal laser endomicroscope.

DETAILED DESCRIPTION:
The gastric mucosal microbiome plays a pivotal role in a series of diseases, such as the H.pylori infection. We hypothesized that mucosal patterns, here visualized by confocal endomicroscopy, may constitute specific microbiome niches.

ELIGIBILITY:
Inclusion criteria:

* Patients scheduled for gastroendoscopy examination
* Aged between 18 and 80 years old

Exclusion criteria:

* Antibiotic, probiotic or prebiotic usage within 2months
* Esophageal, gastric or duodenal cancer or other malignancy
* History of upper GI tract surgery
* Coagulopathy or bleeding disorders
* Allergy to fluorescein sodium
* Pregnant or breast-feeding (for females)
* Impaired renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective patients scheduled for pCLE examination at Qilu Hospital, Shandong University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The operational taxonomy units in gastric mucosal microbiome | 6 months

SECONDARY OUTCOMES:
The diagnostic accuracy of endomicroscopy compared to pathology. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China